CLINICAL TRIAL: NCT05560477
Title: A Prospective, Randomized, Controlled, Double-Blinded, Multi-Center, Phase 1/2b Study to Evaluate the Safety and Efficacy of AM3101 to Augment Meniscal Healing
Brief Title: Study to Evaluate the Safety and Efficacy of AM3101 to Augment Meniscal Healing
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Cincinnati (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency)
Responsible Party: Principal Investigator, Brian Grawe, Principal Investigator, University of Cincinnati
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Protocol Number: SM17091; UC IRB Number: 2019-0468 (Other: University of Cincinnati)
Record Dates: First submitted 2022-09-23; First posted 2022-09-29 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-05

CONDITIONS: Meniscus Tear
Keywords: meniscal repair; complications; morbidities

STUDY DESIGN:
Intervention Model Description: Prospective, randomized, controlled, double-blinded, multi-center study
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: A vial of AM3101 is inverted to mix and aspirated into the barrel of a 5cc syringe in a controlled area to ensure sterility. The saline control will be prepared in a similar fashion. The syringes will be labeled with blinding tape and transferred to the surgical suite.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Treated with repair and AM3101 (Experimental): Syringe containing AM3101 for injection.
  Interventions: Drug: AM3101
- Treated with repair and 0.9% sodium chloride (saline) (Placebo Comparator): Syringe containing commercially available 0.9% sodium chloride for injection.
  Interventions: Drug: Saline Placebo

INTERVENTIONS:
Drug: AM3101 — Injectable drug product.
  Arms: Treated with repair and AM3101
Drug: Saline Placebo — 2 mL 0.9% normal saline
  Arms: Treated with repair and 0.9% sodium chloride (saline)

SUMMARY:
The purpose of this clinical trial is to assess the safety and efficacy of AM3101 to facilitate meniscal repair and reduce the incidence of non-healing complications and morbidities associated with a failed meniscal repair. This is a prospective, randomized, controlled, double-blinded, multi-center study.

DETAILED DESCRIPTION:
Primary Efficacy Objective: Assess the efficacy of AM3101 by evaluating the integrity of repaired meniscal tissue assessed via MRI at 12 months following injection with AM3101 as compared to the integrity of meniscal tissue at 12 months in the control group injected with a saline solution (placebo).

Primary Safety Objective: Assess the safety of AM3101 by evaluating the incidence of individual adverse events and comparing these adverse event rates to incidence rates for the control group injected with a saline solution (placebo).

Secondary Objective: Assess and compare functional outcomes in patients receiving AM3101 following meniscal repair to functional outcomes in the control group injected with a saline solution (placebo).

ELIGIBILITY:
Inclusion Criteria:

1. Male or female ≥ 18 and ≤ 40 years old at time of screening.
2. MRI evidence of ACL plus meniscus tear, or isolated meniscus tear.
3. Body mass index (BMI) ≤ 40 kg/m2.
4. Liver and kidney function panels within normal ranges at time of screening
5. Willing and able to comply with the study procedures and visit schedule, and able to follow oral and written instructions.
6. Willing and able to sign an IRB approved informed consent

Exclusion Criteria:

1. Have any concomitant ligament injury requiring surgical repair or reconstruction other than the ACL.
2. Have a history of previous meniscus injury that currently needs to be treated or has been treated surgically.
3. Have evidence of arthritis ≥ Grade III (Outerbridge classification) in the affected compartment or greater than Kellgren Lawrence Grade 3.
4. Elevated AST or ALT liver enzymes at time of screening
5. Pregnant or nursing mothers, or women planning on getting pregnant during the time they will be participating in the study.
6. Known drug or alcohol dependence currently or within the last year.
7. Participating concurrently in another clinical study or have participated in a clinical study within the last 90 days, or intend to during the course of the study.
8. Any medical condition or other circumstances that might interfere with the ability to return for follow-up visits in the judgment of the Investigator, including any systemic illness, neuromuscular, neurosensory, or musculoskeletal deficiency that would render the subject unable to perform appropriate postoperative rehabilitation.
9. Any condition which, in the judgment of the Investigator, would preclude adequate evaluation of the investigational product's safety and efficacy.
10. Known allergic reaction to simvastatin.
11. Patients currently taking simvastatin, or any other drug that is within the statin drug classification family.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 74 (Estimated)
Dates: Start 2023-04-26 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Healing Assessed via MRI | 12 months
  Presence or absence of healing assessed via MRI
Incidence of Adverse Events | 12 months
  Incidence of adverse events in subjects receiving AM3101 following meniscal repair, as compared to subjects undergoing meniscal repair and injected with a saline solution (placebo).

CONTACTS AND LOCATIONS:
Overall Officials: Brian M Grawe, MD, Principal Investigator — University of Cincinnati
Locations (3):
- United States (3):
  - University of Cincinnati, Cincinnati, Ohio
  - University Hospitals Cleveland Medical Center, Cleveland, Ohio
  - Oregon Health & Science University, Portland, Oregon

IPD SHARING:
Plan to Share IPD: Yes
A public-use version of the dataset will be constructed with contents to be determined by the study PI. Copies of the public-use version of the dataset will be housed at the University of Cincinnati on a secure server along with suitable documentation of this dataset. The public-use version of the dataset will be exported by CRF in one or more files in simple, widely-accessible formats, e.g., .xls, .csv, and/or SAS datasets. Documentation will be in .pdf files.
Supporting Information: Study Protocol, CSR
Time Frame: The public-use version of the database will be made 2 years after the study's main paper is published.
Access Criteria: Outside investigators wishing to conduct analyses using the data will submit a request with objectives, methods, and analysis plan to the PI. Once the request is approved, the public-use version of the dataset, with documentation, will be sent by secure email using e-mail, ftp, or other mutually agreeable transmission method.

REFERENCES:
- [Background] Nepple JJ, Dunn WR, Wright RW. Meniscal repair outcomes at greater than five years: a systematic literature review and meta-analysis. J Bone Joint Surg Am. 2012 Dec 19;94(24):2222-7. doi: 10.2106/JBJS.K.01584. PMID 23318612
- [Background] Xu H, Bouta EM, Wood RW, Schwarz EM, Wang Y, Xing L. Utilization of longitudinal ultrasound to quantify joint soft-tissue changes in a mouse model of posttraumatic osteoarthritis. Bone Res. 2017 Jun 13;5:17012. doi: 10.1038/boneres.2017.12. eCollection 2017. PMID 28638676
- [Background] Proulx ST, Kwok E, You Z, Papuga MO, Beck CA, Shealy DJ, Ritchlin CT, Awad HA, Boyce BF, Xing L, Schwarz EM. Longitudinal assessment of synovial, lymph node, and bone volumes in inflammatory arthritis in mice by in vivo magnetic resonance imaging and microfocal computed tomography. Arthritis Rheum. 2007 Dec;56(12):4024-37. doi: 10.1002/art.23128. PMID 18050199
- [Background] Fukui T, Ii M, Shoji T, Matsumoto T, Mifune Y, Kawakami Y, Akimaru H, Kawamoto A, Kuroda T, Saito T, Tabata Y, Kuroda R, Kurosaka M, Asahara T. Therapeutic effect of local administration of low-dose simvastatin-conjugated gelatin hydrogel for fracture healing. J Bone Miner Res. 2012 May;27(5):1118-31. doi: 10.1002/jbmr.1558. PMID 22275312
- [Background] Oka S, Matsumoto T, Kubo S, Matsushita T, Sasaki H, Nishizawa Y, Matsuzaki T, Saito T, Nishida K, Tabata Y, Kurosaka M, Kuroda R. Local administration of low-dose simvastatin-conjugated gelatin hydrogel for tendon-bone healing in anterior cruciate ligament reconstruction. Tissue Eng Part A. 2013 May;19(9-10):1233-43. doi: 10.1089/ten.TEA.2012.0325. Epub 2013 Jan 14. PMID 23198912
- [Background] Vos LM, Kuijer R, Huddleston Slater JJ, Bulstra SK, Stegenga B. Inflammation is more distinct in temporomandibular joint osteoarthritis compared to the knee joint. J Oral Maxillofac Surg. 2014 Jan;72(1):35-40. doi: 10.1016/j.joms.2013.08.022. Epub 2013 Nov 6. PMID 24210930
- [Background] Donahue RP, Gonzalez-Leon EA, Hu JC, Athanasiou K. Considerations for translation of tissue engineered fibrocartilage from bench to bedside. J Biomech Eng. 2018 Dec 5;141(7):0708021-07080216. doi: 10.1115/1.4042201. Online ahead of print. PMID 30516244
- [Background] Roy TC. Diagnoses and mechanisms of musculoskeletal injuries in an infantry brigade combat team deployed to Afghanistan evaluated by the brigade physical therapist. Mil Med. 2011 Aug;176(8):903-8. doi: 10.7205/milmed-d-11-00006. PMID 21882780
- [Background] Sanders JW, Putnam SD, Frankart C, Frenck RW, Monteville MR, Riddle MS, Rockabrand DM, Sharp TW, Tribble DR. Impact of illness and non-combat injury during Operations Iraqi Freedom and Enduring Freedom (Afghanistan). Am J Trop Med Hyg. 2005 Oct;73(4):713-9. PMID 16222015
- [Background] Hutchinson ID, Moran CJ, Potter HG, Warren RF, Rodeo SA. Restoration of the meniscus: form and function. Am J Sports Med. 2014 Apr;42(4):987-98. doi: 10.1177/0363546513498503. Epub 2013 Aug 12. PMID 23940202
- [Background] Fox AJ, Wanivenhaus F, Burge AJ, Warren RF, Rodeo SA. The human meniscus: a review of anatomy, function, injury, and advances in treatment. Clin Anat. 2015 Mar;28(2):269-87. doi: 10.1002/ca.22456. Epub 2014 Aug 14. PMID 25125315
- [Background] Cox JS, Nye CE, Schaefer WW, Woodstein IJ. The degenerative effects of partial and total resection of the medial meniscus in dogs' knees. Clin Orthop Relat Res. 1975;(109):178-83. doi: 10.1097/00003086-197506000-00026. PMID 1173359
- [Background] Kadam UT, Blagojevic M, Belcher J. Statin use and clinical osteoarthritis in the general population: a longitudinal study. J Gen Intern Med. 2013 Jul;28(7):943-9. doi: 10.1007/s11606-013-2382-8. Epub 2013 Mar 8. PMID 23471638
- [Background] Gupta S, Del Fabbro M, Chang J. The impact of simvastatin intervention on the healing of bone, soft tissue, and TMJ cartilage in dentistry: a systematic review and meta-analysis. Int J Implant Dent. 2019 Apr 9;5(1):17. doi: 10.1186/s40729-019-0168-4. PMID 30963362
- [Background] Zhang S, Matsushita T, Kuroda R, Nishida K, Matsuzaki T, Matsumoto T, Takayama K, Nagai K, Oka S, Tabata Y, Nagamune K, Kurosaka M. Local Administration of Simvastatin Stimulates Healing of an Avascular Meniscus in a Rabbit Model of a Meniscal Defect. Am J Sports Med. 2016 Jul;44(7):1735-43. doi: 10.1177/0363546516638342. Epub 2016 Apr 11. PMID 27159292
- [Background] Zhao BJ, Liu YH. Simvastatin induces the osteogenic differentiation of human periodontal ligament stem cells. Fundam Clin Pharmacol. 2014 Oct;28(5):583-92. doi: 10.1111/fcp.12050. Epub 2013 Nov 8. PMID 24112098
- [Background] Lopez-Alvarez M, Lopez-Puente V, Rodriguez-Valencia C, Angelome PC, Liz-Marzan LM, Serra J, Pastoriza-Santos I, Gonzalez P. Osteogenic effects of simvastatin-loaded mesoporous titania thin films. Biomed Mater. 2018 Feb 2;13(2):025017. doi: 10.1088/1748-605X/aa95f1. PMID 29068320
- [Background] Kramer J, Bartsch M, Krug D, Klinger M, Nitschke M, Rohwedel J. Simvastatin modulates mouse embryonic stem cell-derived chondrogenesis in vitro. Toxicol In Vitro. 2012 Oct;26(7):1170-6. doi: 10.1016/j.tiv.2012.06.013. Epub 2012 Jul 3. PMID 22771337
- [Background] Beck SE, Jung BH, Fiorino A, Gomez J, Rosario ED, Cabrera BL, Huang SC, Chow JY, Carethers JM. Bone morphogenetic protein signaling and growth suppression in colon cancer. Am J Physiol Gastrointest Liver Physiol. 2006 Jul;291(1):G135-45. doi: 10.1152/ajpgi.00482.2005. PMID 16769811
- [Background] Zhang H, Lin CY. Simvastatin stimulates chondrogenic phenotype of intervertebral disc cells partially through BMP-2 pathway. Spine (Phila Pa 1976). 2008 Jul 15;33(16):E525-31. doi: 10.1097/BRS.0b013e31817c561b. PMID 18628692
- [Background] Skottheim IB, Gedde-Dahl A, Hejazifar S, Hoel K, Asberg A. Statin induced myotoxicity: the lactone forms are more potent than the acid forms in human skeletal muscle cells in vitro. Eur J Pharm Sci. 2008 Apr 23;33(4-5):317-25. doi: 10.1016/j.ejps.2007.12.009. Epub 2008 Jan 18. PMID 18294823
- [Background] Crues JV 3rd, Ryu R, Morgan FW. Meniscal pathology. The expanding role of magnetic resonance imaging. Clin Orthop Relat Res. 1990 Mar;(252):80-7. PMID 2406078
- [Background] Schreiner MM, Raudner M, Marlovits S, Bohndorf K, Weber M, Zalaudek M, Rohrich S, Szomolanyi P, Filardo G, Windhager R, Trattnig S. The MOCART (Magnetic Resonance Observation of Cartilage Repair Tissue) 2.0 Knee Score and Atlas. Cartilage. 2021 Dec;13(1_suppl):571S-587S. doi: 10.1177/1947603519865308. Epub 2019 Aug 17. PMID 31422674
- [Background] Marlovits S, Singer P, Zeller P, Mandl I, Haller J, Trattnig S. Magnetic resonance observation of cartilage repair tissue (MOCART) for the evaluation of autologous chondrocyte transplantation: determination of interobserver variability and correlation to clinical outcome after 2 years. Eur J Radiol. 2006 Jan;57(1):16-23. doi: 10.1016/j.ejrad.2005.08.007. Epub 2005 Oct 3. PMID 16203119
- [Background] Trattnig S, Ba-Ssalamah A, Pinker K, Plank C, Vecsei V, Marlovits S. Matrix-based autologous chondrocyte implantation for cartilage repair: noninvasive monitoring by high-resolution magnetic resonance imaging. Magn Reson Imaging. 2005 Sep;23(7):779-87. doi: 10.1016/j.mri.2005.04.010. Epub 2005 Aug 26. PMID 16214608
- [Background] Marlovits S, Striessnig G, Resinger CT, Aldrian SM, Vecsei V, Imhof H, Trattnig S. Definition of pertinent parameters for the evaluation of articular cartilage repair tissue with high-resolution magnetic resonance imaging. Eur J Radiol. 2004 Dec;52(3):310-9. doi: 10.1016/j.ejrad.2004.03.014. PMID 15544911
- [Background] Verdonk P, Dhollander A, Almqvist KF, Verdonk R, Victor J. Treatment of osteochondral lesions in the knee using a cell-free scaffold. Bone Joint J. 2015 Mar;97-B(3):318-23. doi: 10.1302/0301-620X.97B3.34555. PMID 25737514
- [Background] Niemeyer P, Laute V, John T, Becher C, Diehl P, Kolombe T, Fay J, Siebold R, Niks M, Fickert S, Zinser W. The Effect of Cell Dose on the Early Magnetic Resonance Morphological Outcomes of Autologous Cell Implantation for Articular Cartilage Defects in the Knee: A Randomized Clinical Trial. Am J Sports Med. 2016 Aug;44(8):2005-14. doi: 10.1177/0363546516646092. Epub 2016 May 20. PMID 27206690
- [Background] Filardo G, Kon E, Di Martino A, Busacca M, Altadonna G, Marcacci M. Treatment of knee osteochondritis dissecans with a cell-free biomimetic osteochondral scaffold: clinical and imaging evaluation at 2-year follow-up. Am J Sports Med. 2013 Aug;41(8):1786-93. doi: 10.1177/0363546513490658. Epub 2013 Jun 12. PMID 23761684
- [Background] Farr J, Gracitelli GC, Shah N, Chang EY, Gomoll AH. High Failure Rate of a Decellularized Osteochondral Allograft for the Treatment of Cartilage Lesions. Am J Sports Med. 2016 Aug;44(8):2015-22. doi: 10.1177/0363546516645086. Epub 2016 May 13. PMID 27179056
- [Background] Anderson DE, Williams RJ 3rd, DeBerardino TM, Taylor DC, Ma CB, Kane MS, Crawford DC. Magnetic Resonance Imaging Characterization and Clinical Outcomes After NeoCart Surgical Therapy as a Primary Reparative Treatment for Knee Cartilage Injuries. Am J Sports Med. 2017 Mar;45(4):875-883. doi: 10.1177/0363546516677255. Epub 2017 Jan 9. PMID 28068480
- [Background] Aldrian S, Zak L, Wondrasch B, Albrecht C, Stelzeneder B, Binder H, Kovar F, Trattnig S, Marlovits S. Clinical and radiological long-term outcomes after matrix-induced autologous chondrocyte transplantation: a prospective follow-up at a minimum of 10 years. Am J Sports Med. 2014 Nov;42(11):2680-8. doi: 10.1177/0363546514548160. Epub 2014 Sep 9. PMID 25204296
- [Background] Wyatt RW, Inacio MC, Liddle KD, Maletis GB. Factors associated with meniscus repair in patients undergoing anterior cruciate ligament reconstruction. Am J Sports Med. 2013 Dec;41(12):2766-71. doi: 10.1177/0363546513503287. Epub 2013 Sep 12. PMID 24029723
- [Background] Miao Y, Yu JK, Ao YF, Zheng ZZ, Gong X, Leung KK. Diagnostic values of 3 methods for evaluating meniscal healing status after meniscal repair: comparison among second-look arthroscopy, clinical assessment, and magnetic resonance imaging. Am J Sports Med. 2011 Apr;39(4):735-42. doi: 10.1177/0363546510388930. Epub 2011 Jan 10. PMID 21220542
- [Background] Noyes FR, Barber-Westin SD. Long-term Survivorship and Function of Meniscus Transplantation. Am J Sports Med. 2016 Sep;44(9):2330-8. doi: 10.1177/0363546516646375. Epub 2016 May 20. PMID 27206692
- See also: US Food and Drug Administration. Nonclinical review for triamcinolone acetonide (Zilretta) — https://www.accessdata.fda.gov/drugsatfda_docs/nda/2017/208845Orig1s000PharmRedt.pdf
- See also: Merck Sharp & Dohme Corp. Approval package for simvastatin (Zocor). 2011 — https://www.accessdata.fda.gov/drugsatfda_docs/nda/2011/019766s077.pdf
- See also: US Food and Drug Administration. Retrieved on 02 August 2021from — https://www.fda.gov/media/116754/download